CLINICAL TRIAL: NCT04646330
Title: A Phase Ib/II Trial of AK104 Plus Anlotinib in Patients With NSCLC
Brief Title: A Trial of AK104 Plus Anlotinib in NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-208
Record Dates: First submitted 2020-11-23; First posted 2020-11-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK104 10mg/kg Q2W plus anlotinib (Experimental): Subjects receive AK104 10mg/kg every 2-week cycle(Q2W) intravenously (IV) plus anlotinib 1-14days of every 3-week cycle (Q3W) until no more benefits from treatment.
  Interventions: Drug: AK104+anlotinib
- AK104 15mg/kg Q3W plus anlotinib (Experimental): Subjects receive AK104 15mg/kg intravenously (IV) plus anlotinib 1-14days of every 3-week cycle (Q3W) until no more benefits from treatment.
  Interventions: Drug: AK104+anlotinib
- AK104 10mg/kg Q3W plus anlotinib (Experimental): Subjects receive AK104 10mg/kg Q3W plus anlotinib 1-14days of every 3-week cycle until no more benefits from treatment.
  Interventions: Drug: AK104+anlotinib

INTERVENTIONS:
Drug: AK104+anlotinib — Subjects receive AK104 10mg/kg intravenously (IV) every 2-week cycle plus anlotinib on Day 1-14 of every 3-week cycle (Q3W) until progression.
  Arms: AK104 10mg/kg Q2W plus anlotinib
Drug: AK104+anlotinib — Subjects receive AK104 15mg/kg intravenously (IV) every 3-week cycle plus anlotinib on Day 1-14 of every 3-week cycle (Q3W) until progression.
  Arms: AK104 15mg/kg Q3W plus anlotinib
Drug: AK104+anlotinib — Subjects receive AK104 10mg/kg Q3W plus anlotinib 1-14days of every 3-week cycle until progression.
  Arms: AK104 10mg/kg Q3W plus anlotinib

SUMMARY:
This trial is a single arm, two cohorts, phase Ib/II study. All patients are stage IIIB/C or IV NSCLC, Eastern Cooperative Oncology Group (ECOG) performance status 0-1. Cohort 1 includes treatment naïve patients with advanced NSCLC. Cohort 2 includes patients with metastatic or recurrent NSCLC after progression on treatment with PD-1/PD-L1. The primary end point are objective response rate per RECIST1.1 and safety. Secondary end points are progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old (at the time consent is obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Have histologically- or cytologically-confirmed diagnosis of StageIIIB/C or IV NSCLC.
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue obtained from either a core or excisional tumor biopsy.
* Have a life expectancy of at least 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team
* Has adequate organ function as defined by:Absolute neutrophil count ≥ 1,500/µL;Platelets ≥ 100,000/µL;Hemoglobin ≥ 9 g/dL;Crcl ≥ 50ml/min creatinine clearance may be calculated using the institutional/laboratory standard method.Serum total bilirubin ≤ 1.5 x ULN ;Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN ;Albumin ≥28g/L;International Normalized Ratio (INR) and aPTT <1.5 x ULN. Left ventricular ejection fraction ≥50%.
* Have recovered from the effects of any prior radiotherapy or surgery
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Is currently participating in a study of an investigational agent or using an investigational device;
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment;
* Has undergone major surgery within 30 days of Study Day 1;
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases;
* Has carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study;
* Has an active infection requiring systemic therapy;
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator;
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, an average of 1 year
  objective response rate per RECIST1.1

SECONDARY OUTCOMES:
progession-free survival (PFS) | through study completion, an average of 1 year
  progession-free survival per RECIST1.1
overall survival (OS) | through study completion, an average of 1 year
  overall survival per RECIST1.1
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wu, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan cancer hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Chen B, Yao W, Li X, Lin G, Chu Q, Liu H, Du Y, Lin J, Duan H, Wang H, Xiao Z, Sun H, Liu L, Xu L, Xu Y, Xu F, Kong Y, Pu X, Li K, Wang Q, Li J, Li B, Xia Y, Wu L. A phase Ib/II study of cadonilimab (PD-1/CTLA-4 bispecific antibody) plus anlotinib as first-line treatment in patients with advanced non-small cell lung cancer. Br J Cancer. 2024 Feb;130(3):450-456. doi: 10.1038/s41416-023-02519-0. Epub 2023 Dec 18. PMID 38110665